CLINICAL TRIAL: NCT01185067
Title: GRAPe Seed Extract and Ventriculovascular Investigation in Normal Ejection-Fraction Heart Failure
Brief Title: Physiological Effects of Grape Seed Extract in Diastolic Heart Failure
Acronym: GRAPEVINE-HF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Scott L. Hummel, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM00029626
Record Dates: First submitted 2010-08-02; First posted 2010-08-19 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Diastolic Heart Failure; Hypertensive Heart Disease; Heart Failure With Preserved Ejection Fraction; Hypertension; Oxidative Stress
Keywords: Hypertension; Endothelial function; Antioxidants; Oxidative stress; Grapes; Polyphenols; Resveratrol; Quercetin; Anthocyanins; Flavanols; Flavonols; Congestive heart failure; Heart failure with normal ejection fraction; Heart failure with preserved systolic function; HFNEF; HFPSF; HFPEF; DHF
MeSH Terms: conditions — Heart Failure, Diastolic; Hypertension; Heart Failure | interventions — Grape Seed Extract; grp protein, Drosophila; Wine; Polyphenols; Resveratrol; Quercetin; Anthocyanins; Flavonoids; Flavonols; Antioxidants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- grape seed extract capsule (Active Comparator): Grape seed extract (MegaNatural BP, Polyphenolics, Inc.) 300 milligram capsules twice daily for six weeks
  Interventions: Drug: grape seed extract (MegaNatural BP, Polyphenolics, Inc.)
- maltodextrin capsule (Placebo Comparator): Maltodextrin capsules (matched for appearance and taste to grape seed extract capsules) twice daily for six weeks
  Interventions: Drug: grape seed extract (MegaNatural BP, Polyphenolics, Inc.)

INTERVENTIONS:
Drug: grape seed extract (MegaNatural BP, Polyphenolics, Inc.) — Subjects will be randomized in double-blind fashion to either grape seed extract (GSE) or maltodextrin placebo capsules for for 6 weeks. Patient will take 300 mg GSE/placebo twice a day for 6 weeks. Patient will have a 2 week washout period and then cross over to the opposite group for an additional 6 weeks.
  Other Names: grapes; wine; polyphenols; resveratrol; quercetin; anthocyanins; flavonoids; flavanols; flavonols; antioxidants

SUMMARY:
Diastolic heart failure (also known as "heart failure with normal ejection fraction" or "heart failure with preserved ejection fraction") occurs even though the heart muscle's pumping function is normal. In many cases diastolic heart failure is related to stiffening of the heart and blood vessels in people who have high blood pressure. Current guidelines suggest that patients should limit the salt content of their diet, as too much salty food can cause fluid retention and other problems in diastolic heart failure. Studies in animals with diastolic heart failure suggest that antioxidant chemicals found in grapes can block some of the harmful effects of salty diets. Because it is often difficult for patients with diastolic heart failure to maintain a low salt diet, the investigators are researching the effects of the antioxidant properties of grape seed extract, a natural supplement made from grape seeds. The investigators hypothesize that supplementing the diet with grape seed extract (GSE) can decrease the levels of harmful chemicals and improve heart and blood vessel function in patients with diastolic heart failure and a history of high blood pressure.

The University of Michigan research group plans to enroll 25 patients with a history of high blood pressure and diastolic heart failure in a research study. The study will assess the effects of GSE on hormones and other chemicals that can cause heart and blood vessel damage. The investigators will also study the effects of GSE on the ability of the blood vessels and heart muscles to relax at the proper time and speed. Finally, the investigators will observe how GSE affects participants' overall ability to exercise, quality of life, and blood pressure control. Study participants will be randomly assigned to take either GSE or placebo (looks like but does not contain GSE) capsules twice a day for six weeks. After a two-week break, all subjects will cross over to the opposite group of capsules for an additional six-week period. At the start of the study and at the end of each six-week time period study participants will have non-invasive heart and blood vessel testing, blood work and urine tests, and blood pressure monitoring.

ELIGIBILITY:
Inclusion Criteria:

Inclusion:

* Signs and symptoms of heart failure
* Left ventricular ejection fraction ≥ 50% (contrast ventriculography, echocardiography, nuclear scintigraphy, MRI or CT imaging)
* Diastolic dysfunction on previous echocardiogram/catheterization, or indeterminate diastolic function with supporting evidence of heart failure (HF) (as per European Society of Cardiology guidelines)
* History of systemic hypertension
* Age ≥ 50 years
* Willing to adhere to prescribed course of supplementation
* Informed consent

Exclusion Criteria:

* Daily intake of antioxidant supplements or vitamins beyond that provided in a standard daily multivitamin (e.g. high-dose vitamin E or vitamin C)
* NYHA Class IV heart failure symptoms (except during previous hospitalization)
* Hospitalization for decompensated heart failure within past one month
* Severely uncontrolled hypertension (SBP ≥ 180 and.or DBP ≥ 100 at rest, on current antihypertensive regimen
* Uncontrolled diabetes mellitus (hemoglobin A1C > 9%)
* Severe renal (estimated GFR < 30 ml/min) or hepatic disease/failure
* Severe anemia (Hgb < 9)
* Primary exercise limitation due to severe pulmonary disease
* Unacceptably poor echocardiographic images for analysis
* Worse than moderate mitral or aortic stenosis or insufficiency.
* Non-hypertensive cause of HFpEF (e.g. valvular disease, congenital heart disease, amyloidosis, sarcoidosis, constrictive pericardial syndromes)
* Myocardial infarction or unstable angina, including new or worsening anginal syndrome, within the past three months
* Uncontrolled arrhythmia (including non rate-controlled atrial fibrillation)
* Terminal illness expected to result in death within six months or active solid-organ cancer
* Psychiatric disorder (or dementia) with potential to compromise adherence
* Changes in medical regimen for heart disease or hypertension within past 1 month (except diuretic dose adjustment)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2013-11-04 (Actual); Study Completion 2014-02-24 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation (FMD) | Pre-six weeks of investigational drug and placebo intervention
  Ultrasound measure of conduit artery endothelial function
Brachial artery flow-mediated dilation (FMD) | Post-six weeks of investigational drug and placebo intervention
  Ultrasound measure of conduit artery endothelial function

SECONDARY OUTCOMES:
24-hour blood pressure | Pre-six weeks of investigational drug and placebo intervention
  Mean and diurnal variation
EndoPAT arterial endothelial function | Pre-six weeks of investigational drug and placebo intervention
  Plethysmographic measure of resistance arterial endothelial function
Carotid-femoral pulse wave velocity | Pre-six weeks of investigational drug and placebo intervention
Maximal exercise capacity and oxygen consumption | Pre-six weeks of investigational drug and placebo intervention
Resting and post-exercise ventricular systolic and diastolic function | Pre-six weeks of investigational drug and placebo intervention
  Standard and novel echocardiographic measures including strain/strain rate
Urinary 8-isoprostanes | Pre-six weeks of investigational drug and placebo intervention
  Measure of oxidative stress
Heart failure related quality of life | Pre-six weeks of investigational drug and placebo intervention
  Minnesota Living With Heart Failure Questionnaire
24-hour blood pressure | Post-six weeks of investigational drug and placebo intervention
  Mean and diurnal variation
EndoPAT arterial endothelial function | Post-six weeks of investigational drug and placebo intervention
  Plethysmographic measure of resistance arterial endothelial function
Carotid-femoral pulse wave velocity | Post-six weeks of investigational drug and placebo intervention
Maximal exercise capacity and oxygen consumption | Post-six weeks of investigational drug and placebo intervention
Resting and post-exercise ventricular systolic and diastolic function | Post-six weeks of investigational drug and placebo intervention
  Standard and novel echocardiographic measures including strain/strain rate
Urinary 8-isoprostanes | Post-six weeks of investigational drug and placebo intervention
  Measure of oxidative stress
Heart failure related quality of life | Post-six weeks of investigational drug and placebo intervention
  Minnesota Living With Heart Failure Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Scott L Hummel, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Seymour EM, Singer AA, Bennink MR, Parikh RV, Kirakosyan A, Kaufman PB, Bolling SF. Chronic intake of a phytochemical-enriched diet reduces cardiac fibrosis and diastolic dysfunction caused by prolonged salt-sensitive hypertension. J Gerontol A Biol Sci Med Sci. 2008 Oct;63(10):1034-42. doi: 10.1093/gerona/63.10.1034. PMID 18948553
- [Background] Ma L, Gao HQ, Li BY, Ma YB, You BA, Zhang FL. Grape seed proanthocyanidin extracts inhibit vascular cell adhesion molecule expression induced by advanced glycation end products through activation of peroxisome proliferators-activated receptor gamma. J Cardiovasc Pharmacol. 2007 May;49(5):293-8. doi: 10.1097/FJC.0b013e31803c5616. PMID 17513948
- [Background] Sivaprakasapillai B, Edirisinghe I, Randolph J, Steinberg F, Kappagoda T. Effect of grape seed extract on blood pressure in subjects with the metabolic syndrome. Metabolism. 2009 Dec;58(12):1743-6. doi: 10.1016/j.metabol.2009.05.030. Epub 2009 Jul 15. PMID 19608210
- [Background] Kar P, Laight D, Rooprai HK, Shaw KM, Cummings M. Effects of grape seed extract in Type 2 diabetic subjects at high cardiovascular risk: a double blind randomized placebo controlled trial examining metabolic markers, vascular tone, inflammation, oxidative stress and insulin sensitivity. Diabet Med. 2009 May;26(5):526-31. doi: 10.1111/j.1464-5491.2009.02727.x. PMID 19646193